CLINICAL TRIAL: NCT02961309
Title: A Laboratory Model of Increasing THC Potency on Cigarette Smoking
Brief Title: A Laboratory Model of Increasing Delta-9-tetrahydrocannabinol (THC) Potency on Cigarette Smoking
Acronym: MJCIG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BMI-73659
Record Dates: First submitted 2016-11-02; First posted 2016-11-10 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Tobacco Use
Keywords: THC; marijuana; tobacco cigarette; smoking
MeSH Terms: conditions — Tobacco Use; Marijuana Abuse; Smoking | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active THC (Experimental): 5.6% THC via smoked marijuana cigarette
  Interventions: Drug: THC
- Placebo (Experimental): Placebo THC via smoked cigarette
  Interventions: Drug: THC

INTERVENTIONS:
Drug: THC — 1 High-Potency THC (Dosage = 10mg) cigarette (oral smoking) on one day and 1 Placebo on the other day.
  Other Names: marijuana

SUMMARY:
The objective of the proposed research is to investigate how smoking increasing potency of THC (i.e., the psychoactive ingredient in marijuana) changes tobacco cigarette smoking behavior, urges, subjective effects, and abuse liability. This study will be a within-subjects, placebo-controlled study in our clinical laboratory of the effect of active vs. placebo marijuana on cigarette puff topography, exhaled carbon monoxide, urge, subjective effects, and abuse liability among 7 adults who smoke both marijuana and tobacco cigarettes.

DETAILED DESCRIPTION:
The study requires a total of three visits to Battelle's laboratory: one screening visit and two experimental visits. The screening visit will determine eligibility into the study. If eligible, participants will smoke a tobacco cigarette through the Clinical Research Support System (CReSS) puff topography device. Enrolled participants will attend two separate 5-hour experimental visits. Participants will be randomly assigned the order of THC potency (active or placebo), with the assignment blocked by sex. When participants arrive at the laboratory for each visit, they will provide biologic samples to verify compliance with pre-study instructions and then will be taken to a specially ventilated smoking chamber. They will be connected to a continuously-monitoring heart rate and blood pressure machine so that their vital signs can be observed throughout the smoking session. A research assistant will give a marijuana cigarette to the participant. A research assistant will light the cigarette and then exit the room. Participants will follow tape-recorded instructions for smoking the marijuana cigarette through the CReSS device. Upon completion of smoking the marijuana cigarette, participants will complete the Tobacco Craving Questionnaire via paper and pencil and will then be allowed to smoke one of his own tobacco cigarettes through the CReSS puff topography device. Participants will be allowed to smoke as many tobacco cigarettes as they would like for the next 3 hours. Participants will then be given lunch and sent home via taxicab. All participants will receive both potencies (i.e., active and placebo) of marijuana. The active potency of marijuana will be 5.6% THC.

ELIGIBILITY:
Inclusion Criteria:

1. Current US resident;
2. Age ≥ 18 years;
3. Self-reported smoking of marijuana no more than three days per week within the past year;
4. Self-report past-month smoking of marijuana;
5. Self-report daily smoking of at least five cigarettes per day within the past year;
6. Cotinine ≥ 100 ng/mL at the in-person screening visit; and
7. Able to read, understand, and sign informed consent.

Exclusion Criteria:

1. Meets Diagnostic and Statistical Manual-5 (DSM-5) criteria for current (i.e., past year) or past (i.e., lifetime) cannabis use disorder;
2. Meets DSM-5 criteria for any current Axis I disorder, other than tobacco use disorder;
3. Self-reported current desire to stop marijuana or tobacco use, defined as 7 or greater on an 11-rung (scaled of 1-10) Contemplation Ladder for each;
4. Self-reported asthma or chronic obstructive pulmonary disease; and
5. Among females, current pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Puff topography of tobacco cigarette smoked | 30 minutes post-marijuana smoking
  Mean total puff volume

SECONDARY OUTCOMES:
Boost in exhaled breath carbon monoxide after smoking tobacco cigarette | 30 minutes post-marijuana smoking
  Pre- to post-tobacco cigarette smoking difference in exhaled breath carbon monoxide
Self-reported urge to smoke tobacco cigarette | 30 minutes post marijuana smoking
  Pre- to post-tobacco cigarette smoking difference in scores on the Questionnaire of Smoking Urge
Self-reported subjective effects related to tobacco cigarette smoking | 30 minutes post marijuana smoking
  Pre- to post-tobacco cigarette smoking difference in the Nicotine-Drug Effects Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wallace Pickworth, PhD, Principal Investigator — Battelle
Locations (1):
- Battelle Memorial Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No